CLINICAL TRIAL: NCT03503942
Title: The Pre-Diabetes Interventions and Continued Tracking to Ease-out Diabetes (Pre-DICTED) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Ministry of Health, Singapore (Other Government); Health Promotion Board, Singapore (Other Government); Singapore Clinical Research Institute (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREDICTED2017
Record Dates: First submitted 2017-10-13; First posted 2018-04-20 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Participants in the treatment arm will receive structured group-based lifestyle interventions with stepwise addition of metformin for selected high-risk participants.
  Interventions: Behavioral: Lifestyle modification; Drug: Metformin; Other: Financial incentives
- Control (No Intervention): Participants in the control arm will receive the current standard of care for pre-diabetes which includes counseling on lifestyle modifications and follow up by primary care physicians.

INTERVENTIONS:
Behavioral: Lifestyle modification — Participants in the treatment arm will receive structured, locally tailored, group-based lifestyle interventions that consist of a core intervention phase (3 months) and a maintenance phase (33 months). The core intervention phase will consist of twice weekly group sessions on nutrition, exercise and goal-setting within the first 6 weeks followed by 6 weeks of self-directed lifestyle modification. During the maintenance phase, the participants will receive monthly short message service (SMS) on health tips as well as 6 monthly telephone calls from program coordinators.
  Arms: Treatment arm
Drug: Metformin — Metformin will be will be prescribed to treatment group participants at highest risk of diabetes conversion (i.e.IFG + IGT or IFG + HbA1c ≥6.0%) after at least 6 months of lifestyle interventions at a starting dose of 250 mg twice a day followed by up-titration to 500 mg twice a day after 3 months if the participants do not experience any gastrointestinal side effects.
  Arms: Treatment arm
Other: Financial incentives — Participants will be given cash incentives if they meet the weight loss target, which is pre-defined as 5% of baseline weight, at the 3rd, 6th, 12th, 18th, 24th, 30th and 36th month of study period.
  Arms: Treatment arm

SUMMARY:
The Pre-DICTED (Pre-Diabetes Intervention and Continued Tracking to Ease-out Diabetes) program is a community-based diabetes prevention program. This study aims to test the effectiveness of structured, group-based lifestyle interventions with stepwise addition of metformin, if required, among subjects with pre-diabetes in multi-ethnic Singapore.

DETAILED DESCRIPTION:
The Pre-DICTED program is designed as a randomized, controlled, pragmatic trial. The program targets to recruit up to 846 overweight/obese (BMI ≥23.0) adults (age 18-64) with isolated impaired fasting glucose (IFG), isolated impaired glucose tolerance (IGT), or IFG + IGT in Singapore. The follow-up period will be 3 years.

Eligible subjects will be identified through community, primary care clinics and hospital-based diabetes screening program. Following informed consent, eligible participants will be randomised into the control or the treatment arm.

Participants in the control arm will receive the current standard of care for pre-diabetes which includes counseling on lifestyle modifications and follow up by primary care physicians.

Participants in the treatment arm will undergo a 3-month, locally tailored, group-based lifestyle intervention program (consisting of nutrition workshops, exercise sessions and goal-setting workshop) plus subsequent stepwise addition of metformin for selected participants at the highest risk of progression to diabetes at ≥ 6 months of follow-up. Financial incentives will be awarded to participants who achieve weight lost of ≥5% of baseline weight during follow-up period.

The primary outcome of diabetes incidence will be assessed bi-annually and compared across the study arms. Secondary outcomes will include weight, waist circumference, fasting plasma glucose (FPG), 2-h glucose, HbA1c, physical activity, diet and metformin adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Singapore citizens or permanent residents
2. Age between 18 and 64
3. Body mass index (BMI) ≥ 23.0 kg/m2
4. Pre-diabetes diagnosed based on:

   1. fasting plasma glucose 6.1 - 6.9 mmol/L (Impaired fasting glucose; IFG) and/or
   2. 2-hr plasma glucose in 75g oral glucose tolerance test (OGTT) 7.8 - 11.0 mmol/L (Impaired glucose tolerance; IGT) (Laboratory tests to be done within 6 months of enrolment)

Exclusion Criteria:

1. Individuals with diabetes mellitus
2. Health conditions impeding participation in lifestyle change programme (e.g. active cancer, recent myocardial event within 6 months, heart failure, chronic kidney disease)
3. Current pregnancy or breast feeding
4. Treatment with medications known to alter glucose tolerance
5. Known allergic reaction to metformin

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 751 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Diabetes incidence | 3 years
  The primary outcome, diabetes incidence, will be diagnosed based on a single, annual OGTT or the semi-annual FPG (Fasting plasma glucose) test

SECONDARY OUTCOMES:
Weight | 3 years
  Weight in kg
Waist circumference | 3 years
  Waist circumference in cm
HbA1c | 3 years
  HbA1c in %
Fasting plasma glucose | 3 years
  Fasting plasma glucose in mmol/L
2-hour plasma glucose | 3 years
  2-hour plasma glucose post oral glucose challenge in mmol/L
International physical activity questionnaire (IPAQ) score | 3 years
  IPAQ score in MET minutes a week
Metformin adherence | Up to 30 months
  Metformin adherence assessed by pill counts

CONTACTS AND LOCATIONS:
Overall Officials: Yong Mong Bee, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung KF, Gandhi M, Lam AYR, Julianty S, Chia AYM, Tan GCS, Goh SY, Ho ETL, Koh AFY, Tan GSW, Shum EJW, Finkelstein EA, Jafar TH, Teoh YL, van Dam RM, Whitton C, Thumboo J, Bee YM. The Pre-Diabetes Interventions and Continued Tracking to Ease-out Diabetes (Pre-DICTED) program: study protocol for a randomized controlled trial. Trials. 2021 Aug 6;22(1):522. doi: 10.1186/s13063-021-05500-5. PMID 34362409